CLINICAL TRIAL: NCT00138424
Title: A Randomized, Placebo-Controlled, Dose-Escalation Study to Assess the Safety and Effect of Cidofovir in Renal Transplant Recipients With BK Virus Nephropathy
Brief Title: Cidofovir in Renal Transplant Recipients With BKVN
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-047; CASG 209
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2011-04

CONDITIONS: BK Virus (Nephropathy)
Keywords: Vistide®, Cidofovir, renal transplant, BK Virus Nephropathy
MeSH Terms: conditions — Kidney Diseases | interventions — Cidofovir

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Cidofovir (Experimental): 32 subjects will be randomized to 1 of 3 possible cohorts. Cohort I will receive dose 0.25 mg/kg; Cohort II will receive 0.5 mg/kg, Cohort III will receive 1.0 mg/kg. Maximum tolerated dose is to be determined.
  Interventions: Drug: Cidofovir
- Placebo (Placebo Comparator): 16 subjects to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cidofovir — Cidofovir is a marketed product for treatment of Cytomegalovirus disease (retinitis) in human immunodeficiency virus (HIV) infected patients. It is packaged as a sterile, hypertonic aqueous solution for intravenous infusion only. Dosages: 0.25 mg/kg, 0.5 mg/kg, and 1.0 mg/kg.
  Arms: Cidofovir
Drug: Placebo — The control for this study is sterile, 0.9% normal saline for intravenous use.
  Arms: Placebo

SUMMARY:
This study will look at the safety, tolerability and effectiveness of cidofovir in kidney transplant patients who have been diagnosed with BK virus nephropathy (BKVN), a viral condition that can cause patients to reject transplanted kidneys. Up to 48 adult (age 18 years and older) kidney or pancreas transplant recipients with newly diagnosed BKVN will receive 1 of 3 cidofovir dose levels or placebo (non medicated substance) to identify the maximum tolerated dose. Dosing will be administered intravenously (by a tube running into a blood vessel). In addition to the screening visit, volunteers will actively participate for approximately 8-10 weeks with a single follow up phone call at 4 months. Blood samples, urine samples, eye exams and physical exams are included in study procedures.

DETAILED DESCRIPTION:
The primary objectives of this randomized, double-blind, placebo-controlled, dose-escalation study are to evaluate the safety and tolerability of 3 dose levels of cidofovir when administered to renal transplant recipients with BK virus nephropathy and to identify the maximum tolerated doses (MTD) among the 3 dose levels of cidofovir in renal transplant recipients with BK virus nephropathy. The secondary study objectives are to evaluate the antiviral effect of cidofovir at each of 3 dose levels; to evaluate the pharmacokinetics (PK) of cidofovir in renal transplant recipients with underlying renal impairment; to evaluate the pharmacodynamics (PD) of cidofovir in this setting; to evaluate allograft function at the completion of the study; and to assess allograft rejection at the completion of the study. Patients with BKVN (virus nephropathy) diagnosed by positive plasma polymerase chain reaction (PCR) or renal allograft biopsy will be randomized to receive study drug within 60 days of the date of the renal biopsy or plasma PCR assay that established the diagnosis of BKVN. The study consists of three dose cohorts (0.25 mg/kg, 0.5 mg/kg and 1.0 mg/kg); each cohort will consist of approximately 12 subjects randomized 2:1 to receive either cidofovir or placebo (0.9% normal saline) to define the MTD among the three specified doses of cidofovir. Once the MTD is established, approximately 12 additional patients will be enrolled at that dose. The MTD is defined as the dose in which no more than 2 of the 8 cidofovir treated subjects experience a dose limiting toxicity (DLT). The target enrollment is 48 subjects if all dose cohorts are fully enrolled. A 25% over-enrollment may be tolerated to allow for continued enrollment of subjects in the lower dose cohort if data are under concomitant review by the Data and Safety Monitoring Board (DSMB) or to replace non-evaluable study participants. Study participants who have been randomized and have received cidofovir/placebo (in any cohort) will be considered non-evaluable if they discontinue from the study or die for any reason except toxicities definitely related to study treatment, including DLTs. These subjects may be replaced. There will be a 5-week drug administration period (4 doses) followed by a 2 week end-of-study observation and evaluation period for each cohort. At about 3 months after last dose of study infusion, a member of the research staff will assess the study participant and counsel on pregnancy status via a phone call. The study will be overseen by a DSMB who will review the data after each dose cohort is completed. The primary endpoint of the study will assess the safety and tolerability of cidofovir in kidney transplant recipients this will be assessed by enumeration of adverse events (AEs) reported by the subjects and/or investigator, and changes observed in the physical examination (including vital signs) and laboratory evaluations during the drug administration and end-of-treatment observation and evaluation periods. The severity and relationship of AEs to receipt of study drug will be determined because the primary endpoint is focusing on the safety. The secondary endpoints are the effect of cidofovir on BK virus as determined by: percentage of subjects who achieve an undetectable BK virus urine and plasma PCR between baseline and end of treatment; rate of reduction in urine and plasma BK virus load by quantitative PCR between baseline and end of treatment; and time to reduction in BK virus urine and plasma PCR; the detailed PK of cidofovir will be evaluated in subjects at the MTD; the PD of cidofovir will be assessed by quantitating the change in BK virus deoxyribonucleic aci

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to 18 years.
* Kidney or kidney/pancreas transplant recipient.
* New onset BK Virus Nephropathy (BKVN) diagnosed by a positive plasma polymerase chain reaction (PCR) assay for BK virus deoxyribonucleic acid (DNA) or by a renal biopsy demonstrating BK virus (by immunohistochemistry, electron microscopy and/or in situ hybridization) obtained as part of standard medical care within 60 days prior to receipt of first dose of study drug.
* BK virus load in plasma greater than 10,000 copies/mL within prior 21 days.
* Glomerular filtration rate greater than 30 mL/min using Levey calculations.
* Absolute neutrophil count greater than 1000/microliter [with granulocyte colony stimulating factor (GCSF) support as necessary].
* Women must be post-menopausal, surgically sterile or willing to use adequate contraception (barrier method with spermicide, intrauterine device, oral contraceptives, implant or other licensed hormone method) from time of study enrollment through 1 month after the last dose of study treatment. Men must be surgically sterile or willing to use contraception (barrier method with spermicide) from time of study enrollment through 3 months after the last dose of study treatment.

Exclusion Criteria:

* Unable to provide valid informed consent.
* History of intolerance to cidofovir or related compounds (i.e. other nucleotide derivatives [adefovir or tenofovir]).
* Pregnant or breast feeding women.
* Prior treatment with cidofovir within the last 2 weeks.
* Receipt of another investigational drug with proven nephrotoxic drug interaction with cidofovir or known antipolyoma virus activity one month prior to study entry.
* Contraindication to renal biopsy (e.g., anticoagulant medication, unwilling to undergo biopsy).
* Currently receiving or anticipated to receive any of the following within 2 weeks of randomization:
* Amphotericin preparation (intravenous)
* Aminoglycosides (intravenous)
* Platinum - based chemotherapeutic agents
* NSAIDs - non steroidal anti-inflammatory drugs (aspirin given for cardioprotective treatment is acceptable up to 650 mg per oral daily)
* Foscarnet
* Pentamidine (intravenous)
* Probenecid
* Leflunomide
* Hypotony or uveitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-05; Primary Completion 2010-06 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Alabama Hospital - Nephrology, Birmingham, Alabama
  - California Pacific Medical Center - Sutter Pacific Medical Foundation - Transplant Nephrology, San Francisco, California
  - University of California San Francisco Medical Center at Parnassus - Organ Transplant, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Northwestern University - Comprehensive Transplant Center, Chicago, Illinois
  - The University of Chicago Medical Center - Kindney Trasnplant - Nephrology, Chicago, Illinois
  - University of Minnesota Medical Center, Fairview - Infectious Diseases and International Medicine, Minneapolis, Minnesota
  - Mayo Clinic, Rochester - Infectious Diseases, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center - Infectious Disease, Lebanon, New Hampshire
  - Dallas Nephrology Associates - Dallas Transplant Institute, Dallas, Texas
  - University of Washington - Medicine, Seattle, Washington
  - University of Wisconsin Hospital and Clinics - Clinical Science Center - Nephrology, Madison, Wisconsin

REFERENCES:
- [Derived] Razonable RR. Management of viral infections in solid organ transplant recipients. Expert Rev Anti Infect Ther. 2011 Jun;9(6):685-700. doi: 10.1586/eri.11.43. PMID 21692673

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort I - Cidofovir; Cohort I - Placebo: One dose (0.25 mg/kg/week-days 0, 7, 21, 35, 49)
- Cohort II - Cidofovir; Cohort II - Placebo: One dose (0.5 mg/kg/week-days 0, 7, 21, 35, 49)
Period: Overall Study
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Started | 9 | 5 | 5 | 3
Completed | 9 | 4 | 5 | 3
Not Completed | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo | Total
Number analyzed (Participants) | 9 | 5 | 5 | 3 | 22
Age, Customized [Number; unit: participants]
  < 30 years old | 1 | 2 | 0 | 0 | 3
  30-39 years old | 0 | 0 | 0 | 0 | 0
  40-49 years old | 1 | 2 | 0 | 1 | 4
  50-59 years old | 3 | 1 | 2 | 0 | 6
  60-69 years old | 4 | 0 | 2 | 1 | 7
  >= 70 years old | 0 | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 0 | 4
  Male | 6 | 4 | 5 | 3 | 18
Region of Enrollment [Number; unit: participants]
  United States | 9 | 5 | 5 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Cidofovir Assessed by Enumeration of Adverse Events Per Subject
Description: The measure is the number of adverse events (ie: events that are change from baseline)experienced by subjects. The median or average number of events and the range of events across all subjects is reported.
Time Frame: Baseline through day 49
Measure: Median (Full Range); unit: Event
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Event | 3 [2 to 15] | 4 [1 to 4] | 3 [3 to 5] | 7 [2 to 11]

2. Secondary Outcome: The Effect of Cidofovir on BK Virus Determined by Percentage of Subjects Achieving an Undetectable BK Virus in Urine and Plasma PCR
Description: The outcome measure is the percent of subjects that achieved non-detectable BK virus in the urine and plasma polymerase chain reaction (PCR) at day 35 after staring study drug. Undetectable is a PCR viral load of less than 200.
Time Frame: Day 35.
Population: Percentage of subjects
Measure: Number; unit: percentage of subjects
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
percentage of subjects
  Plasma | 0 | 20 | 0 | 0
  Urine | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage Change of Viral Load in Urine and Plasma BK Virus by Quantitative PCR Between Baseline and Each Visit
Description: The percent change in viral load from baseline to day 7, day 21 and day 49 as measured in the urine and measured in the blood. A drop is identified by use of '-', an increase in viral load has no sign in front of the number.
Time Frame: Baseline, and each visit: day 7, 21, 35 and 49.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Percent Change
  Day 7 Plasma | 21.6 [-195.2 to 60.7] | 61.9 [-17.3 to 99.8] | 21.2 [2.5 to 70.1] | 7.9 [-268.8 to 36.1]
  Day 7 Urine | 9.1 [-149.3 to 87.9] | 19.1 [-55299.7 to 80.0] | -3.1 [-319.5 to 26.5] | 1.6 [-579.6 to 26.4]
  Day 21 Plasma | 35.9 [-387.5 to 88.1] | 75.6 [-75.6 to 99.8] | 58.4 [-6.3 to 89.4] | 53.9 [-174.9 to 71.9]
  Day 21 Urine | 18.3 [-3.7 to 99.6] | 26.2 [-108553.1 to 94.5] | 8.1 [-102.1 to 60.1] | 11.1 [-63.6 to 97.4]
  Day 35 Plasma | 44.8 [-295.2 to 93.3] | 91.3 [2.7 to 99.8] | 76.2 [35.9 to 93.2] | 83.3 [-402.0 to 93.8]
  Day 35 Urine | 27.6 [-32.1 to 99.7] | 29.9 [-88968.7 to 97.8] | 25.5 [3.2 to 76.8] | 8.3 [-7.1 to 92.4]
  Day 49 Plasma | 56.5 [-22.8 to 96.5] | 95.0 [-72.4 to 99.6] | 76.7 [15.8 to 91.3] | 65.1 [-1094.4 to 75.5]
  Day 49 Urine | 42.4 [-142.3 to 99.8] | 86.1 [-65494.3 to 95.8] | -0.7 [-31.1 to 86.5] | 12.9 [-51.5 to 86.4]

4. Secondary Outcome: Subjects Achieving 50% Reduction Viral Load in Plasma and Urine
Time Frame: Baseline through day 49.
Measure: Number; unit: Participants
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Participants
  Number of Subjects at 50% Reduction in Plasma | 6 | 4 | 5 | 2
  Number of Subject at 50% Reduction in Urine | 4 | 3 | 2 | 1

5. Secondary Outcome: Number of Days to at Least 50% Reduction of Viral Load in Plasma and Urine
Time Frame: Baseline through day 49.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Days
  Plasma | 21.5 [7 to 51] | 7.5 [7 to 21] | 22 [7 to 50] | 20.5 [20 to 21]
  Urine | 14.5 [7 to 21] | 35 [7 to 49] | 29 [22 to 36] | 20 [20 to 20]

6. Primary Outcome: Number of Adverse Events by Grade of Event
Description: Adverse events are reported as grades:
  Toxicity Grade I: a mild event (an event that requires minimal or no treatment and does not interfere with the subject's daily activities.
  Toxicity Grade II: a moderate event (an event that results in a low level of inconvenience or concern with the therapeutic measures and may cause some interference with functioning.
  Toxicity Grade III: a severe event (an event that interrupts a subject's usual daily activity and may require systemic drug therapy or other treatment and may be incapacitating.
  Toxicity Grade IV: Life threatening (any adverse drug experience that places the patient or subject at immediate risk of death from the reaction as it occurred)
Time Frame: Baseline through day 49.
Measure: Number; unit: Events
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Events
  Grade 1 | 26 | 4 | 10 | 2
  Grade 2 | 2 | 6 | 1 | 2
  Grad3 3 | 0 | 2 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Related Adverse Events
Description: The investigator's assessment of an AE's relationship to study drug is part of the documentation process. All adverse events had their relationship to study product assessed using the following terms: associated (related)or not associated (not related). To help assess, the following guidelines were used.
  * Associated - There was a known temporal relationship and/or, if re-challenge was done, the event abates with de-challenge and reappears with re-challenge and/or the event was known to occur in association study product or with a product in a similar class of study products
  * Not Associated -the AE was completely independent of study product administration; and/or evidence existed that the event was definitely related to another etiology.
Time Frame: Baseline through day 49.
Population: Number of Related Events
Measure: Number; unit: Events
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Events | 6 | 6 | 1 | 1

8. Primary Outcome: Changes Observed in the Physical Examination : Respiratory Rate (Per Minute)
Description: Respiratory rate is the number of breaths per minute.
Time Frame: Baseline through day 49.
Population: subjects whose respiratory rate was measured at baseline visit and at day 49 visit.
Measure: Median (Full Range); unit: Change in Breaths per Minute
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Change in Breaths per Minute | 0 [-4 to 6] | 0 [-4 to 2] | 0 [-4 to 2] | -2 [-4 to 0]

9. Primary Outcome: Changes Observed in the Physical Examination: Blood Pressure (mm/hg)
Description: Blood pressure (BP) is the pressure exerted by circulating blood upon the walls of blood vessels. "Blood pressure" usually refers to the arterial pressure of the systemic circulation. During each heartbeat, blood pressure varies between a maximum (systolic) and a minimum (diastolic) pressure. The measure is the difference between the baseline systolic and baseline diastolic value with the day 49 systolic and day 49 diastolic value.
Time Frame: Baseline through day 49.
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
mm Hg
  Systolic Blood Pressure | 10 [-31 to 38] | -4 [-8 to 51] | -3 [-17 to 39] | 3 [-46 to 6]
  Diastolic Blood Pressure | 1 [-14 to 1] | 6 [2 to 14] | 10 [-8 to 22] | -4 [-25 to 2]

10. Secondary Outcome: Allograft Function at the Completion of the Study
Description: Glomerular filtration rate (GFR) is a test used to check how well the kidneys are working. Specifically, it estimates how much blood passes through the tiny filters in the kidneys, called glomeruli, each minute. The normal health GFR is about 90 - 120 mL/min/1.73 m2. Older people will have lower normal GFR levels, because GFR decreases with age.
  Abnormal Results are expected to be below 60 mL/min/1.73 m2 for 3 or more months are a sign of chronic kidney disease. A GFR result below 15 mL/min/1.73 m2 may be a sign of kidney failure.
Time Frame: Day 49.
Population: subjects that had GFR at each visit last visit
Measure: Median (Full Range); unit: mL/min/1.73 m2
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
mL/min/1.73 m2 | 42.7 [26.5 to 72.9] | 40.3 [30.0 to 57.8] | 45.1 [36.1 to 90.5] | 63.2 [22.6 to 84.7]

11. Secondary Outcome: Allograft Rejection.
Description: Allograft rejection is the number of subjects that rejected their kidney by the end of the study.
Time Frame: Day 49.
Population: Number of rejections
Measure: Number; unit: Participants
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Participants | 0 | 0 | 0 | 0

12. Primary Outcome: Changes Observed in the Physical Examination: Body Temperature (Fahrenheit)
Description: The temperature is a measure of body temperature in fahrenheit (F). The measure is a change between baseline temperature and day 49 temperature.
Time Frame: Baseline through day 49.
Population: Subject's last visit minus baseline visit
Measure: Median (Full Range); unit: Temperature (F)
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Temperature (F) | 0.18 [-1.82 to 0.18] | 0.72 [-0.54 to 60.46] | -0.42 [-1 to 0.5] | 0.3 [-0.7 to 4.3]

13. Primary Outcome: Changes Observed in the Physical Examination: Heart Rate (Per Minute)
Description: The heart rate is the number of heart beats per minute. The outcome measure is the change from baseline heart rate to day 49 heart rate.
Time Frame: Baseline through day 49.
Population: Subject's whose heart rate was measured at baseline and day 49 visit
Measure: Median (Full Range); unit: Change in Beats per Minute
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Change in Beats per Minute | -3 [-22 to 1] | 3 [-17 to 13] | 4 [-14 to 21] | -4 [-7 to 48]

14. Primary Outcome: Number of Subjects Experiencing at Least One Laboratory Abnormality
Description: The following lab values assessed during the 49 days of subject involvement were the following: hemoglobin, hematocrit, platelets, sodium, potassium, chloride, bicarbonate, blood urea nitrogen (BUN), serum creatinine, calcium, phosphorous, serum albumin, glucose, uric acid, magnesium, total protein, total bilirubin, alanine aminotransferase (ALT), asparate aminotransferase (AST) and alkaline phosphate. The outcome measure is the number of subjects experiencing at least 1 grade 1 (mild) or higher event.
Time Frame: Baseline through day 49
Measure: Number; unit: Participants
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Number analyzed (Participants) | 9 | 5 | 5 | 3
Participants
  WBC | 3 | 3 | 1 | 0
  Hemoglobin | 6 | 5 | 4 | 2
  Hematocrit | 6 | 5 | 2 | 3
  Platelets | 3 | 2 | 3 | 1
  Sodium | 3 | 2 | 0 | 2
  Potassium | 1 | 1 | 1 | 0
  Chloride | 4 | 5 | 3 | 1
  Bicarbonate | 5 | 3 | 2 | 2
  BUN | 9 | 5 | 4 | 2
  Serum Creatinine | 8 | 5 | 4 | 3
  Calcium | 5 | 0 | 2 | 1
  Phosphorous | 5 | 2 | 1 | 0
  Serum Albumin | 4 | 1 | 1 | 2
  Glucose | 7 | 2 | 3 | 1
  Uric Acid | 1 | 2 | 0 | 0
  Magnesium | 5 | 2 | 2 | 1
  Total Protein | 4 | 3 | 0 | 1
  Total Bilirubin | 2 | 0 | 0 | 1
  ALT (SGPT) | 3 | 0 | 0 | 0
  AST (SGOT) | 2 | 3 | 0 | 1
  Alkaline Phosphate | 4 | 0 | 2 | 0

15. Secondary Outcome: The Pharmacodynamics of Cidofovir Will be Assessed by Correlating the Percent Change in BK Virus DNA in Urine and Plasma With Pharmacokinetic Changes Between Baseline Through Day 35
Description: PK parameter change from baseline to day 35 for Cmax.
Time Frame: Baseline through day 35
Measure: Median (Full Range); unit: ng/mL
Groups:
- Cohort I - Cidofovir: One dose (0.25 mg/kg/week - days 0, 7, 21, 35, 49)
- Cohort II - Cidofovir: One dose (0.5 mg/kg/week - days 0, 7, 21, 35, 49)
Arm/Group | Cohort I - Cidofovir | Cohort II - Cidofovir
Number analyzed (Participants) | 9 | 5
ng/mL | 190.4 [-212.2 to 5173.9] | -233.9 [-338.3 to 242.9]
Statistical Analysis 1: Comparison: Cohort I - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in plasma vs the PK Cmax parameter; Test type: Superiority or Other; p = 0.57, Spearman Correlation; Spearman Correlation = 0.24
Statistical Analysis 2: Comparison: Cohort I - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in urine vs the PK Cmax parameter; Test type: Superiority or Other; p = 0.53, Spearman Correlation; Spearman Correlation = 0.26
Statistical Analysis 3: Comparison: Cohort II - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in plasma vs the PK Cmax parameter; Test type: Superiority or Other; p = 0.62, Spearman Correlation; Spearman Correlation = -0.30
Statistical Analysis 4: Comparison: Cohort II - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in urine vs the PK Cmax parameter; Test type: Superiority or Other; p = 0.10, Spearman Correlation; Spearman Correlation = 0.80

16. Secondary Outcome: The Pharmacodynamics of Cidofovir Will be Assessed by Correlating the Percent Change in BK Virus DNA in Urine and Plasma With Pharmacokinetic Changes Between Baseline and Day 35
Description: PK parameter change from baseline to day 35 for AUC4 and AUC12
Time Frame: Baseline through day 35
Measure: Median (Full Range); unit: hr*mg/L
Arm/Group | Cohort I - Cidofovir | Cohort II - Cidofovir
Number analyzed (Participants) | 9 | 5
hr*mg/L
  AUC4 | 0.5 [-0.5 to 3.9] | -0.1 [-0.5 to 0.8]
  AUC12 | 0.3 [-0.7 to 4.2] | 0.1 [-0.5 to 1.5]
Statistical Analysis 1: Comparison: Cohort I - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in plasma vs the PK AUC4 parameter; Test type: Superiority or Other; p = 0.87, Spearman Correlation; Spearman Correlation = 0.07
Statistical Analysis 2: Comparison: Cohort I - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in urine vs the PK AUC4 parameter; Test type: Superiority or Other; p = 0.46, Spearman Correlation; Spearman Correlation = 0.31
Statistical Analysis 3: Comparison: Cohort II - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in plasma vs the PK AUC4 parameter; Test type: Superiority or Other; p = 0.49, Spearman Correlation; Spearman Correlation = -0.41
Statistical Analysis 4: Comparison: Cohort II - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in urine vs the PK AUC4 parameter; Test type: Superiority or Other; p = 0.05, Spearman Correlation; Spearman Correlation = 0.87
Statistical Analysis 5: Comparison: Cohort I - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in plasma vs the PK AUC12 parameter; Test type: Superiority or Other; p = 0.78, Spearman Correlation; Spearman Correlation = 0.12
Statistical Analysis 6: Comparison: Cohort I - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in urine vs the PK AUC12 parameter; Test type: Superiority or Other; p = 0.18, Spearman Correlation; Spearman Correlation = 0.52
Statistical Analysis 7: Comparison: Cohort II - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in plasma vs the PK AUC12 parameter; Test type: Superiority or Other; p = 0.75, Spearman Correlation; Spearman Correlation = 0.20
Statistical Analysis 8: Comparison: Cohort II - Cidofovir; Spearman correlation co-efficient utilized to determine viral load changes in urine vs the PK AUC12 parameter; Test type: Superiority or Other; p = 0.75, Spearman Correlation; Spearman Correlation = 0.20

ADVERSE EVENTS:
Time Frame: SAEs were reported within one business day of awareness of the event by completing Serious Adverse Event Report. Events were reported from start of study drug use to end of study..
Arm/Group | Cohort I - Cidofovir | Cohort I - Placebo | Cohort II - Cidofovir | Cohort II - Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/5 | 0/5 | 1/3
Other Adverse Events (participants affected / at risk) | 6/9 | 4/5 | 3/5 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I - Cidofovir (N=9) | Cohort I - Placebo (N=5) | Cohort II - Cidofovir (N=5) | Cohort II - Placebo (N=3)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transplant Rejection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I - Cidofovir (N=9) | Cohort I - Placebo (N=5) | Cohort II - Cidofovir (N=5) | Cohort II - Placebo (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye burns (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transplant Rejection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study closed early due to failure to enroll in a timely manner.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less